CLINICAL TRIAL: NCT03802799
Title: An Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of ZYN002 Administered as a Transdermal Gel to Children, Adolescents, and Young Adults With Fragile X Syndrome
Brief Title: Open Label Extension to Assess the Long-Term Safety and Tolerability of ZYN002 in Children and Adolescents With FXS
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zynerba Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYN2-CL-017
Record Dates: First submitted 2018-12-26; First posted 2019-01-14 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-02

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZYN002 (Experimental): ZYN002 - cannabidiol Transdermal Gel
  Interventions: Drug: ZYN002 - Cannabidiol Transdermal Gel

INTERVENTIONS:
Drug: ZYN002 - Cannabidiol Transdermal Gel — Pharmaceutically manufactured. Cannabidiol formulated as a clear gel (transdermal delivery)
  Other Names: Cannabidiol Transdermal Gel

SUMMARY:
ZYN002 is a pharmaceutically manufactured Cannabidiol that is developed as a clear gel that can be applied to the skin (called transdermal delivery).

The gel will be applied to clean, dry, intact skin of the shoulders and/or upper arms.

Participants from the ZYN2-CL-016 and ZYN2-CL-033 studies who meet the inclusion criteria and none of the exclusion criteria for study ZYN2-CL-017 are eligible.

Parents/caregivers will apply the study gel twice daily for the 52-week treatment period.

DETAILED DESCRIPTION:
This is an open-label extension, multiple-center study, to assess the long-term safety and tolerability of cannabidiol administered as ZYN002, a transdermal gel, for the treatment of child and adolescent patients with Fragile X Syndrome (FXS). Male and female patients with FXS will be treated for up to 72 months. Up to 450 male and female patients, ages 3 to 18 years will be enrolled.

Parents/caregivers will apply the study gel twice daily for the 52-week treatment period.

Participants from study ZYN-CL-016 who weigh less than or equal to 35 kg, will receive 1 sachet of ZYN002, applied every 12 hours (± 2 hours).

Participants from study ZYN-CL-016 who weigh more than 35 kg will receive 2 sachets of ZYN002, applied every 12 hours (± 2 hours).

Participants from study ZYN-CL-033 who weigh less than or equal to 30 kg, will receive 1 sachet of ZYN002, applied every 12 hours (± 2 hours).

Participants from study ZYN-CL-033 who weigh more than 30 kg will receive 2 sachets of ZYN002, applied every 12 hours (± 2 hours).

Participants from study ZYN-CL-033 who weigh more than 50 kg will receive 3 sachets of ZYN002, applied every 12 hours (± 2 hours).

At the Investigator's discretion, the dose may be increased or decreased at any time after the first month of treatment (for example due to weight changes during the course of the study).

Participants who are taking anti-epileptic drugs may have an additional one or two weeks of treatment after the 52 week treatment period to taper off study treatment.

Blood samples will be collected for safety analysis of ZYN002. Additionally, the parents/caregivers will be asked to complete some questionnaires. There will be other questionnaires and scales that will be completed at the site by the study doctor and/or with the participant and their parents/caregivers.

Patients that complete Month 12 will be allowed to continue for another 12 months of treatment if they qualify. Patients will be evaluated again annually at Months 24 and 36, and 48 in order to remain in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participated in study ZYN2-CL-016 or Study ZYN2-CL-033.
* Patients and parents/caregivers agree to abide by all study restrictions and comply with all study procedures.
* Patients and parents/caregivers must be adequately informed of the nature, risks of the study, and give written informed consent prior to enrollment in ZYN2-CL-017.
* In the Investigator's opinion, the patients and parents/caregivers are reliable and are willing and able to comply with all protocol requirements and procedures.
* Females of childbearing potential must have a negative pregnancy test at all designated visits

Exclusion Criteria:

* Patient is receiving any investigational drugs (not ZYN002) or using any experimental devices.
* Patient has an ongoing serious adverse event (SAE) or has experienced a SAE in ZYN2-CL-016 or ZYN2-CL-033, which in the opinion of the Investigator, should exclude them from participation.
* Females who are pregnant, nursing, or planning a pregnancy; females of childbearing potential and male patients with a partner of childbearing potential who are unwilling or unable to use an acceptable method of contraception for the duration of therapy and for three months after the last dose of trial drug.
* Patients who have alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels ≥ 2 times the upper limit of normal (ULN) or has alkaline phosphatase levels ≥ 3 times the ULN as determined from patient safety laboratories.

Ages: 3 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 550 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety and tolerability of ZYN002 administered as a transdermal gel formulation. | Up to 96 month.
  Safety assessment will include collection of any treatment emergent adverse events

SECONDARY OUTCOMES:
To evaluate the long-term efficacy of ZYN002 in the treatment of symptoms of FXS. | Change from baseline to end of treatment
  Change from Baseline (last assessment prior to the first dose of ZYN002) in the ABC-CFXS subscale scores.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (19):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Science 37, Culver City, California
  - Amnova Clinical Research, LLC, Irvine, California
  - UC Davis Health System, MIND Institute, Sacramento, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Han Phan, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Masonic Institute of Developing Brain, Minneapolis, Minnesota
  - University of Mississipi Medical Center, Jackson, Mississippi
  - The Fragile X Spectrum Disorder Clinic at Icahn School of Medicine at Mount Sinai, Division of Medical Genetics, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - Primary Children's Hospital, Salt Lake City, Utah
- Australia (3):
  - Westmead Children's Hospital, Sydney, New South Wales
  - Lady Cilento Children's Hospital - South Brisbane, Brisbane, Queensland
  - Genetics Clinics Australia, Melbourne, Victoria
- Wellington Hospital, Wellington, New Zealand
- United Kingdom (3):
  - Research Space, Leicester, Leicestershire
  - Children's Clinical Research Facility, Royal Hospital for Children and Young People, Edinburgh, Lothian
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry-Kravis E, Hagerman R, Cohen J, Budimirovic D, Buchanan CB, Silove N, Tich N, Thibodeau A, Dobbins T, Sebree T, O'Quinn S, Albers DS, Bzdek KG, Nomikos G, Budur K. Long-term safety and tolerability of transdermal cannabidiol gel in children and adolescents with Fragile X syndrome (ZYN2-CL-017): an interim analysis of an ongoing open-label extension study. J Neurodev Disord. 2025 Nov 18;17(1):69. doi: 10.1186/s11689-025-09657-x. PMID 41254489
- [Derived] Heussler HS. Emerging Therapies and challenges for individuals with Angelman syndrome. Curr Opin Psychiatry. 2021 Mar 1;34(2):123-128. doi: 10.1097/YCO.0000000000000674. PMID 33395098